CLINICAL TRIAL: NCT04273516
Title: Aspirin Plus Rivaroxaban Efficacy and Safety in Embolic Stroke of Undetermined Source: A Randomized, Placebo Controlled, Outcome Assessor Blind, Feasibility Study
Brief Title: Rivaroxaban Plus ASA in Embolic Stroke of Undetermined Source(AREST-ESUS)
Acronym: AREST-ESUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant Professor in Neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3498
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Prevention
Keywords: ESUS; DOACS; Prevention
MeSH Terms: conditions — Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Tablet Rivaroxaban 2.5 mg 2 times daily plus ASA 80 mg daily
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet
- Comparator (Placebo Comparator): Tab ASA 80 mg daily plus placebo ( similar to rivaroxaban tablet) 2 times daily
  Interventions: Drug: Rivaroxaban placebo tablets

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — Tablet Rivaroxaban 2.5 mg 2 times daily add to standard treatment ASA 80 mg daily
  Other Names: Axabin 2.5
  Arms: Intervention
Drug: Rivaroxaban placebo tablets — Placebo tablets add to ASA 80 mg daily that is standard treatment
  Other Names: Placebo
  Arms: Comparator

SUMMARY:
Approximately 17% of all patients with stroke are classified as having ESUS, which is associated with a considerable rate of stroke recurrence 4-5 % per year.

Despite recent scientific advances in acute ischemic stroke treatment in recent decades,consensus treatment of all guidelines is still ASA

DETAILED DESCRIPTION:
This is an outcome assessor blind, randomized, parallel, placebo-controlled pilot study on ischemic stroke of undetermined source which will be conducted in Bu Ali Sina hospital in Sari, Iran.

Patients with recent stroke with criteria of ESUS, will be randomized to Rivaroxaban 2.5 mg BID plus ASA 80 mg daily or ASA 80 mg plus placebo (1:1 ratio) and have visit every 3 month until 1 year

ELIGIBILITY:
Inclusion Criteria:

1. signing the inform consent
2. recent ischemic stroke ( 7-60) days with criteria of ESUS
3. only one risk factors of potential embolic source including:

   1. PTFV1 in standard ECG ≥0.05 mm.s or ≥0.005 mv.s
   2. LVH in standard ECG( Sokolow index≥ 35 mm) or on echocardiography
   3. Moderate or severe valvular disorder on echocardiography (except MS)
   4. PFO without indication of occlusion
   5. Left atrium enlargement in echocardiography

Exclusion Criteria:

1. History of hypersensitivity to the investigational medicinal product
2. Indication for anticoagulation
3. Indication for dual antiplatelet therapy
4. Contraindication to investigational medications
5. History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
6. Gastrointestinal bleed or major surgery within 3 months
7. Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
8. HAS-BLED score >3
9. Severe non-cardiovascular comorbidity with life expectancy < 3 months
10. Severe renal failure, defined as Glomerular Filtration Rate (GFR) <15ml/min, Dialysis, transplant, Cr >2.26 mg/dL
11. Severe hepatic insufficiency, Cirrhosis or Bilirubin >2x Normal or AST/ALT/AP >3x Normal
12. Modified Rankin Scale of >=4 at time of randomization or inability to swallow medications.
13. Hemorrhagic transformation of infarction detected by Brain CT or MRI at the time of drug application
14. Radiological or microbiological evidence of COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of stroke recurrence | Rate of stroke recurrence during one year fallow up
  Number of stroke events during 1 year of study
Rate of major bleeding | During 1 year of study
  Rate of major bleeding according to criteria of the International Society of Thrombosis and Hemostasis

SECONDARY OUTCOMES:
Rate of stroke or systemic embolisms | During 1 year of study
  Number of stroke or systemic embolisms recurrence during 1 year of study
Mortality rate | During 1year of study
  Number of all cause mortality during study
Rate of non-major bleeding | During 1year of study
  Rate of non-major bleeding according to criteria of the International Society of Thrombosis and Hemostasis
Rate of intracranial bleeding | During 1year of study
  Rate of ICH during study
Rate of fatal bleeding | During 1 year of study
  Rate of fatal bleeding in any site

CONTACTS AND LOCATIONS:
Overall Officials: Athena Sharifi-Razvi, Principal Investigator — mazandaran university of medical science; Monireh Ghazaeian, Study Director — mazandaran university of medical science
Locations (1):
- Bou- Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Data will be available for researchers and scientific persons after request and review the proposal .